CLINICAL TRIAL: NCT04600388
Title: Retrospective, Observational Survey Study to Assess the Efficacy and Safety of Nerivio for the Acute Treatment of Menstrual Migraine
Brief Title: Efficacy and Safety of Nerivio for the Acute Treatment of Menstrual Migraine
Status: Completed | Type: Observational
Sponsor: Theranica (Industry)
Responsible Party: Sponsor
Other Study IDs: TCH009
Record Dates: First submitted 2020-10-19; First posted 2020-10-23 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-10

CONDITIONS: Menstrual Migraine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Nerivio — Nerivio Remote Electrical Neuromodulation (REN) device

SUMMARY:
Post-marketing, retrospective, observational survey study. Users (menstruating women only) of Nerivio who have used Nerivio at least 4 times between October 2019 and December 2020 will be contacted by email and/or through an app notification and will be asked to complete a 5-minute online anonymous survey assessing satisfaction, effectiveness, and safety. Eligible users will sign an informed consent form (the consent language will appear as the first page of the survey, and participants will click either "agree" or "disagree" to the consent statement; those who click "agree" will proceed to the survey, those who click "disagree" will be brought to an exit page) and complete a survey asking about their satisfaction with Nerivio and the effectiveness and safety of the device for acute treatment of menstrual migraine. During the survey, participants will be screened to verify that they have menstrual migraine (self-reported) and have used Nerivio to treat menstrual migraines.

DETAILED DESCRIPTION:
This study aims to evaluate the safety and efficacy of Nerivio for the acute treatment of menstrual migraine (pure menstrual migraine or menstrually-related migraine).

Up to 500 US-based adults aged 18-55 years old who have been prescribed the Nerivio device and have used it at least 4 times between October 2019 and December 2020.

Informed consent must be obtained from the participant before any protocol-related activities are performed. The consent language will appear as the first page of the survey, and participants will click either "agree" or "disagree" to the consent statement; those who click "agree" will proceed to the survey, those who click "disagree" will be brought to an exit page.

Users of Nerivio whose details are in the sponsor's database will be contacted by email (provided by the patient during the sign-up process in the Nerivio app required to use the device) and/or through an app notification and will be asked to complete a 5-minute online survey assessing satisfaction, effectiveness, and safety. Participants will sign an informed consent form which will appear as the first page of the survey using open-ended questions, multiple choice questions and Likert scales. Participants will be directed to provide honest opinions regarding the device use for menstrual migraine. No additional information will be collected, and no medical records will be used in this investigation.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18-55 years
2. Participants have used Nerivio at least 4 times
3. Participants experience menstrual migraines (pure menstrual migraine or menstrually-related migraine; self-reported)
4. Participants have used Nerivio to treat menstrual migraine

Exclusion Criteria:

1. Non-menstruating women

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Menstrual migraine is female only
Study Population: Menstruating women aged 18-55 years who have used Nerivio at least 4 times and have menstrual migraine.
Sampling Method: Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-11-10 (Actual)

PRIMARY OUTCOMES:
Efficacy of Nerivio during menstrual migraines | 3 months
  Efficacy of Nerivio for headache relief during menstrual migraines rated on a 5-point Likert scale (1 - Not at all effective, 2 - Slightly effective, 3 - Moderately effective, 4 - Very effective, 5- Extremely effective)
Satisfection of using Nerivio during menstrual migraines | 3 months
  Satisfection of using Nerivio during menstrual migraines rated on a 5-point Likert scale )1 - Not at all satisfied, 2 - Slightly dissatisfied, 3 - Neutral, 4 - Slightly satisfied, 5 -Extremely satisfied)

SECONDARY OUTCOMES:
Mean headache relief | 3 months
  Mean percentage of menstrual migraine attacks in which relief was achieved
Medication consumption | 3 months
  Percentage of menstrual migraine attacks in which acute medication was avoided following using the Nerivio
Reduction of menstrual cramps | 3 months
  Percentage of patients reports reduction in menstrual cramps following using of Nerivio

CONTACTS AND LOCATIONS:
Overall Officials: Hida Nierenburg, MD, Principal Investigator — Nuvance Health
Locations (1):
- Vassar Ambulatory Surgical Center, Poughkeepsie, New York, United States

IPD SHARING:
Plan to Share IPD: No
No plean for IPD

REFERENCES:
- [Derived] Nierenburg H, Rabany L, Lin T, Sharon R, Harris D, Ironi A, Wright P, Chuang L. Remote Electrical Neuromodulation (REN) for the Acute Treatment of Menstrual Migraine: a Retrospective Survey Study of Effectiveness and Tolerability. Pain Ther. 2021 Dec;10(2):1245-1253. doi: 10.1007/s40122-021-00276-7. Epub 2021 Jun 17. PMID 34138449